CLINICAL TRIAL: NCT01873859
Title: Incidence of Lactic Acidosis After Coronary Angiography and Angioplasty in Diabetic Patients on Continued Metformin Therapy With Normal Renal Function.
Brief Title: Safety of Continuing Metformin in Diabetic Patients With Normal Kidney Function Receiving Contrast Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Saeed Alipour Parsa, Alipour Parsa S., Assistant professor of cardiology, Cardiovascular Research Center, Modarres hospital, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: sbcvrc-43-891128
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus; Lactic Acidosis
Keywords: Lactic acidosis; Contrast media; Angiography; Diabetic; Metformin
MeSH Terms: conditions — Diabetes Mellitus; Acidosis, Lactic | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- On-metformin (Active Comparator): Diabetic patients receiving contrast media without discontinuing metformin.
  Interventions: Drug: Metformin
- Off-metformin (No Intervention): Diabetic patients receiving contrast media with discontinuation of metformin.

INTERVENTIONS:
Drug: Metformin — Incidence of lactic acidosis in diabetic patients receiving contrast media in the presence of metformin.
  Other Names: Glucophage
  Arms: On-metformin

SUMMARY:
The purpose of this study is to determine whether metformin causes lactic acidosis in diabetic patients with preserved kidney function, undergoing coronary angiography or angioplasty with new contrast media.

In other words is it necessary to discontinue metformin before these procedures, even when Iodixanol is used as contrast media, which is isosmolar agent and much more safer than urografin which was the main agent in the previous studies that were the base of present guidelines?

DETAILED DESCRIPTION:
Although metformin is not directly nephrotoxic, it has been postulated that can impair gluconeogenesis from lactate, which may lead to lactate accumulation under circumstances such as acute renal failure. In diabetic patients receiving metformin, this condition can be encountered in the setting of acute renal failure following contrast media administration, during coronary angiography i.e. contrast-induced nephropathy. As a result, it has been a part of routine clinical practice to discontinue metformin before angiography to prevent metformin-associated lactic acidosis (MALA). However, there is no general consensus regarding the incidence of MALA and evidence for such intervention is poor. On the other hand, discontinuation of metformin can be associated with detrimental effects on glycemic control and thereby may increase cardiovascular risk in diabetic patients undergoing percutaneous coronary interventions. Consequently, questions have been raised recently regarding the routine discontinuation of metformin, in low-risk patients undergoing coronary angiography.

The present study was designed to assess the role of metformin in lactate production in a group of diabetic patients with normal renal function; and to address the questions about significance of routine discontinuation of metformin in low risk patients undergoing coronary angiography.

Iodixanol will be the only contrast media in all patients, because of its low nephrotoxicity. Serum blood urea nitrogen and creatinin; as well as arterial blood gases will be evaluated prior to angiography, and repeated 24 and 48 hours after the procedure. Glomerular filtration rate (GFR) is calculated using Cockcroft-Gault formula {GFR= 0.85 (for women)}.

Contrast-induced acute kidney injury is defined as a 25-50% or 0.3-0.5 mg/dl net increase in creatinine concentration compared to the baseline values. Metformin-associated lactic acidosis (MALA) is defined as an arterial pH (potential of hydrogen)<7.35 and plasma lactate concentration >5 mmol⁄L. In the M (-) group metformin will re-started 48 hours after angiography, albeit in the absence of evidence of lactic acidosis and GFR of >60 mL/min per 1.73 m2.

A written informed consent is taken from all participants and institutional review board has already approved the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients receiving metformin who were scheduled for:

  * coronary angiography
  * coronary angioplasty

Exclusion Criteria:

* Patients who had contraindication for metformin administration, such as:

  * decompensated heart failure
  * severe liver disease
  * severe hypoxemia
  * GFR<60 mL/min per 1.73 m2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Alipour Parsa, Principal Investigator — Cardiovascular research center, Modarres hospital, Shahid Beheshti University of Medical Sciences
Locations (1):
- Cardiovascular research center, Modarres hospital., Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Goergen SK, Rumbold G, Compton G, Harris C. Systematic review of current guidelines, and their evidence base, on risk of lactic acidosis after administration of contrast medium for patients receiving metformin. Radiology. 2010 Jan;254(1):261-9. doi: 10.1148/radiol.09090690. PMID 20032157

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | On-metformin | Off-metformin
Started | 83 | 83
Completed | 83 | 79
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: 166 metformin consumping patients were enrolled. Patients were randomly allocated to continue metformin during peri-angiography period or to stop the medication 24 hours prior the procedure. Four patients in the M (-) group did not complete the study protocol and were excluded from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | On-metformin | Off-metformin | Total
Number analyzed (Participants) | 83 | 79 | 162
Age, Continuous [Mean (Full Range); unit: years] | 61.57 [41 to 84] | 60.1 [41 to 76] | 60.9 [41 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 40 | 83
  Male | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Lactic Acidosis
Description: Metformin-associated lactic acidosis (MALA) was defined as an arterial pH <7.35 and plasma lactate concentration >5 mmol ⁄ L.
Time Frame: 48 hrs
Measure: Number; unit: participants
Arm/Group | On-metformin | Off-metformin
Number analyzed (Participants) | 83 | 79
participants | 0 | 0

2. Primary Outcome: Change of Baseline Creatinine 48 hr After Recieving Contrast Media in the Presence or Absence of Metformin Use.
Time Frame: 48 hours from the baseline
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- On-metformin: Diabetic patients receiving contrast media without discontinuing metformin.
  Metformin: rise of creatinin 48 hr after recieving contrast media.
Arm/Group | On-metformin | Off-metformin
Number analyzed (Participants) | 83 | 79
mg/dl | 1.05 (0.116) | 0.99 (0.159)

ADVERSE EVENTS:
Arm/Group | On-metformin | Off-metformin
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/79
Other Adverse Events (participants affected / at risk) | 0/83 | 0/79

LIMITATIONS AND CAVEATS:
unable to follow patient's creatinine and acidosis for more than 48 hr.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes